CLINICAL TRIAL: NCT03021967
Title: Preliminary Study: Perceptions of Doctors and Caregivers Confronted With Adult Patients in Advanced or Terminal Stage of a Severe, Progressive and Incurable Pathology in the Services of the Hospitals University of Strasbourg Including Beds Identified Palliative Care
Brief Title: Perceptions of Health Professionals Confronted With Palliative Situations
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5581
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Incurable Pathologies
Keywords: incurable pathologies; palliative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Hospitals, doctors and caregivers, who take care of increasingly heavy patients, are faced with ever more complex situations, particularly in the case of severe, progressive, and incurable pathologies.

Thanks to their willingness and expertise, these care providers try to guarantee the continuity and quality of care for both patients and patients in a palliative situation. Nevertheless, these same actors testify to the complexity they encounter in the care of patients in advanced or terminal stages, especially since the concept of "palliative care", which was often erroneously reduced during the Any end of life and therefore death, remains a source of questions, contradictions, even resistances.

In this context, how do physicians and caregivers appropriate palliative care? How do they react to the complexity and intensity of certain situations? Do they have specific expectations of help or support in the face of certain difficulties? Are there actions to be carried out and developed to make the aid given to these actors of the palliative approach more efficient?

These are the topics that the HUS palliative care service proposes to explore through a study of physicians and caregivers working in HUS services for adult patients with LISP.

ELIGIBILITY:
Inclusion Criteria:

* Major hospitals, doctors and caregivers, who take care of increasingly heavy patients

Exclusion Criteria:

* Patient under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals, doctors and caregivers, who take care of increasingly heavy patients,
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent CALVEL, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service Soins Palliatifs, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No